CLINICAL TRIAL: NCT00490451
Title: A Phase 2 Study of LY573636-Sodium Administered as Second-line or Third-line Treatment in Patients With Unresectable or Metastatic Soft Tissue Sarcoma
Brief Title: A Study of LY573636-Sodium in the Treatment of Patients With Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10408; H8K-MC-JZAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Results first posted 2018-05-02 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — N-((5-bromo-2-thienyl)sulfonyl)-2,4-dichlorobenzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY573636 (Experimental)
  Interventions: Drug: LY573636-sodium

INTERVENTIONS:
Drug: LY573636-sodium — LY573636 dose is dependent on patient's height, weight, and gender to target a specific maximum concentration (Cmax). LY573636 is administered intravenously every 21 or 28 days until disease progression or other criteria for patient discontinuation are met.
  Other Names: Tasisulam

SUMMARY:
The primary purpose of the study is to estimate the time from the first dose of LY573636-sodium (hereafter referred to as LY573636) to the date your physician determines that your disease has progressed or worsened.

DETAILED DESCRIPTION:
Patients will receive a 2-hour intravenous infusion of study drug (LY573636) once every 21 days or 28 days depending on their target dose. Radiological imaging scans will be performed before the first dose of study drug and then after every other treatment. Patients will be assessed for clinical progression at every visit and for response approximately every 42 days or 56 days (every other cycle).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of soft tissue sarcoma that is unresectable or metastatic
* Have received one or two (but no more than two) prior treatment regimens for metastatic soft tissue sarcoma, one of which must have included doxorubicin (adriamycin).
* Must have stopped all previous treatments for cancer, including chemotherapy, radiation therapy or other investigational treatments for cancer for at least 30 days

Exclusion Criteria:

* Participants with primary bone sarcoma (for example osteosarcoma, Ewing's sarcoma, chondrosarcoma), gastrointestinal stromal tumor (GIST) and Kaposi's sarcoma
* Serious pre-existing medical problems (as determined by your doctor)
* Have received more than two previous systemic treatment regimens for unresectable or metastatic soft tissue sarcoma
* Have a second primary cancer (unless cancer-free for more than 2 years)
* Active treatment with Warfarin (Coumadin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires, Argentina
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Ryan CW, Matias C, Agulnik M, Lopez-Pousa A, Williams C, de Alwis DP, Kaiser C, Miller MA, Ermisch S, Ilaria R Jr, Keohan ML. A phase II study of tasisulam sodium (LY573636 sodium) as second-line or third-line treatment for patients with unresectable or metastatic soft tissue sarcoma. Invest New Drugs. 2013 Feb;31(1):145-51. doi: 10.1007/s10637-012-9819-5. Epub 2012 Apr 27. PMID 22539091
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- LY573636 Target Cmax 420 µg/mL: LY573636 dose is dependent on participant's height, weight, and gender to target maximum concentration (Cmax) of 420 micrograms/milliliter (µg/mL) and is administered intravenously every 21- or 28-day cycle until disease progression or other criteria for participant discontinuation are met.
- LY573636 Target Cmax 360 µg/mL: LY573636 dose is dependent on participant's height, weight, and gender to target maximum concentration (Cmax) of 360 micrograms/milliliter (µg/mL) and is administered intravenously every 21- or 28-day cycle until disease progression or other criteria for participant discontinuation are met.
Period: Overall Study
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 360 µg/mL
Started | 63 | 38
Completed | 0 | 0
Not Completed | 63 | 38
Not completed — Adverse Event | 3 | 3
Not completed — Death | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Investigator Decision | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Progressive Disease | 53 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 360 µg/mL | Total
Number analyzed (Participants) | 63 | 38 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (15.29) | 52.6 (13.57) | 53.3 (14.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 21 | 51
  Male | 33 | 17 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 3 | 2 | 5
  Caucasian | 54 | 29 | 83
  East Asian | 0 | 2 | 2
  Hispanic | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 30 | 73
  Argentina | 11 | 4 | 15
  Spain | 9 | 4 | 13
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Classifies participants according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  Participants
    0 - Fully active | 30 | 18 | 48
    1 - Ambulatory, restricted strenuous activity | 33 | 19 | 52
    Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Defined as the time from date of first dose to the first observation of progression of disease (PD) or death due to any cause. PD was determined using the Response Evaluation Criteria In Solid Tumors (RECIST) criteria (version 1.0). PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion.
Time Frame: First treatment dose to measured progressive disease or death from any cause up to 15.57 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 360 µg/mL
Number analyzed (Participants) | 63 | 38
months | 2.64 [1.41 to 3.38] | 1.38 [1.38 to 1.54]

2. Secondary Outcome: Percentage of Participants With Complete Response or Partial Response (Objective Response Rate)
Description: Objective response rate is the percentage of participants with complete response (CR) or partial response (PR), as assessed according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines (version 1.0). CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. Objective response rate is calculated as a total number of participants with CR or PR divided by the total number of participants treated multiplied by 100.
Time Frame: First treatment dose to measured progressive disease or death due to any cause up to 15.57 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 360 µg/mL
Number analyzed (Participants) | 63 | 38
percentage of participants
  Complete Response (CR) | 0.0 [NA to NA] — No participants had complete response (CR), therefore 90% confidence interval is not available. | 0.0 [NA to NA] — No participants had complete response (CR), therefore 90% confidence interval is not available.
  Partial Response (PR) | 3.2 [0.0 to 6.8] | 2.6 [0.0 to 6.9]

3. Secondary Outcome: Percentage of Participants With Complete Response (CR), Partial Response (PR), or Stable Disease (SD) (Clinical Benefit Rate)
Description: Clinical Benefit Rate = (CR + PR + SD)/N as classified according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines (version 1.0), where N = total number of participants with at least one dose of study drug. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: First treatment dose to measured progressive disease or death due to any cause up to 15.57 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 360 µg/mL
Number analyzed (Participants) | 63 | 38
percentage of participants | 46.0 [35.7 to 56.4] | 26.3 [14.6 to 38.1]

4. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY573636
Time Frame: Predose up to 2 hours postdose in Cycles 1 and 2 (21- or 28-day cycle)
Population: Participants who received study drug and had pharmacokinetic (PK) data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 360 µg/mL
Number analyzed (Participants) | 62 | 33
micrograms/milliliter (µg/mL)
  Cycle 1 | 386.0 (14.0) | 325.7 (14.5)
  Cycle 2: number analyzed (Participants) | 51 | 28
  Cycle 2 | 346.5 (15.0) | 351.8 (12.8)

5. Secondary Outcome: Overall Survival Time
Description: Defined as the time from date of first dose to the date of death due to any cause.
Time Frame: First treatment dose to death due to any cause up to 26.51 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 360 µg/mL
Number analyzed (Participants) | 63 | 38
months | 8.71 [7.39 to 16.23] | 12.25 [7.79 to 15.64]

6. Secondary Outcome: Duration of Overall Objective Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression of disease or death due to any cause. CR or PR is classified according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines (version 1.0). CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions.
Time Frame: Time of response to progressive disease or death up to 15.57 months
Population: Zero participants analyzed. Duration of Response for CR and PR data was not collected for analysis due to N=0 CR and N=3 PR.
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 360 µg/mL
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Duration of Stable Disease (SD)
Description: Duration of SD is defined from date of documented SD or better to first date of progression of disease (PD) (assessed every other cycle during study therapy, or every 2 months during post-therapy until PD). SD is neither sufficient shrinkage to qualify for partial response (PR) nor sufficient increase to qualify for PD. PR is ≥30% decrease in sum of longest diameter of target lesions. PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion.
Time Frame: Time from documented SD or better to first date of progressive disease up to 15.57 months
Population: All enrolled participants who received at least 1 dose of study drug and had a best overall response of stable disease or better.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 360 µg/mL
Number analyzed (Participants) | 29 | 10
months | 4.44 [4.14 to 5.42] | 5.91 [2.76 to 7.89]

8. Secondary Outcome: Number of Participants With Adverse Events (Safety)
Description: Data are presented as number of participants who experienced serious adverse events or all other nonserious adverse events during the study. A summary of serious adverse events and other nonserious adverse events is located in the Reported Adverse Event section.
Time Frame: First treatment dose up to 26.51 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 360 µg/mL
Number analyzed (Participants) | 63 | 38
Participants
  Serious Adverse Events | 23 | 10
  Other Nonserious Adverse Events | 59 | 36

ADVERSE EVENTS:
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 360 µg/mL
Serious Adverse Events (participants affected / at risk) | 23/63 | 10/38
Other Adverse Events (participants affected / at risk) | 59/63 | 36/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY573636 Target Cmax 420 µg/mL (N=63) | LY573636 Target Cmax 360 µg/mL (N=38)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 3 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (7) | 4 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY573636 Target Cmax 420 µg/mL (N=63) | LY573636 Target Cmax 360 µg/mL (N=38)
Anaemia (Blood and lymphatic system disorders) | 19 (27) | 6 (11)
Leukopenia (Blood and lymphatic system disorders) | 20 (26) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 14 (15) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 15 (27) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 21 (37) | 8 (15)
Palpitations (Cardiac disorders) | 3 (3) | 2 (2)
Tachycardia (Cardiac disorders) | 3 (3) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 10 (12) | 5 (6)
Constipation (Gastrointestinal disorders) | 17 (17) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 17 (22) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (12) | 7 (7)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 6 (11) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (6) | 4 (5)
Asthenia (General disorders) | 4 (5) | 3 (3)
Chest discomfort (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 25 (27) | 9 (9)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 2 (3) | 2 (2)
Mucosal inflammation (General disorders) | 5 (5) | 4 (4)
Oedema peripheral (General disorders) | 12 (12) | 4 (4)
Pain (General disorders) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 7 (7) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 (5) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 5 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 1 (1)
Weight decreased (Investigations) | 8 (8) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (9) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 (13) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (23) | 6 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 7 (10) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 5 (5) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 5 (5) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6) | 2 (2)
Anxiety (Psychiatric disorders) | 6 (6) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (8) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days